CLINICAL TRIAL: NCT05028439
Title: Endoscopic Radiofrequency Ablation Combined With Gemcitabine and S-1 in Paitiens for Unresectable Cholangiocarcinoma：A Randomized Open-label Clinical Trial
Brief Title: RFA Combined With Chemotherapy for Unresectable Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Hangzhou Cancer Hospital (Other); Changhai Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Director, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-08-17
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cholangiocarcinoma
Keywords: biliary tract cancer; radiofrequency ablation; S-1; Gemcitabine
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAF combined with gemcitabine and S-1 group (Experimental): Patients will receive endobiliary radiofrequency ablation ( RFA) followed by plastic stent(s) placement, and be treated with gemcitabine and S-1 within 1 month after RFA.
  Interventions: Device: radiofrequency ablation; Drug: Chemotherapy drug
- RFA-only gruop (Placebo Comparator): Patients will only receive endobiliary radiofrequency ablation ( RFA) followed by plastic stent(s) placement
  Interventions: Device: radiofrequency ablation

INTERVENTIONS:
Device: radiofrequency ablation — All patients underwent biliary sphincterotomy. Cholangiogram was performed to confirm stricture location, length and diameter. The Habib Endo HPB (Hepatobiliary) probe (EMcision, HitchinHerts, UK) was then advanced over a wire at the level of the biliary stricture and ablation using ERBE generator set at 7-10 watts for a time period of 90-120 s was conducted. A 1- to 2-min resting period after energy delivery was allowed before moving the catheter along the length of the stricture to ablate the rest of the stricture. Plastic stent(s) were placed after RFA depending on the location of the malignant obstruction
Drug: Chemotherapy drug — Gemcitabine 1 000 mg/m2 intravenously on day 1，8; S-1 80 mg/m2 was taken orally twice for two weeks. The curative effect was evaluated comprehensively for each 2 cycles of chemotherapy
  Other Names: oral fluoropyrimidine
  Arms: RAF combined with gemcitabine and S-1 group

SUMMARY:
Extrahepatic cholangiocarcinoma is a malignant tumor that is highly malignant and difficult to diagnose and treat early. Endobiliary radiofrequency ablation (RFA) has been reported to be a beneficial treatment option for palliation of malignant biliary strictures. Within the bile duct, RFA appears to be safe and may result in decreased tumor ingrowth. To date, little is known about the role of the addition of systemic chemotherapy to RFA for cholangiocarcinoma. The aim of this study is to compare the efficacy and safety of RAF combined with Gemcitabine and S-1 in patients with unresectable cholangiocarcinoma.

DETAILED DESCRIPTION:
Over 60 % of common bile duct (CBD) obstructions are due to malignancy, and the majority of neoplasms are unresectable at the time of diagnosis. Biliary drainage with placement of metal or plastic stents for palliation is the therapy of choice in this set of patients.

Radiofrequency ablation (RFA) is well established method for treatment of some solid tumors, like liver cancer, lung cancer, etc. Recently, an endoscopically applicable radiofrequency probe, HabibTM EndoHBP catheter, was approved for clinical use. RFA uses a high-frequency alternating current to generate heat and achieve coagulative necrosis when in contact with tissue. Many studies showed RFA with biliary stent was a beneficial treatment option for palliation of malignant biliary strictures. However, most of therapeutic effects were expected to delay bile duct obstruction rather than to decrease the tumor. Recently orally available chemotherapeutic agent, S-1, an oral fluoropyrimidine, was reported as effective in patients with bile duct adenocarcinoma. To date, little is known about the role of the addition of systemic chemotherapy to RFA for cholangiocarcinoma.

The aim of this study is to compare the efficacy and safety of RAF combined with Gemcitabine and S-1 in patients with unresectable cholangiocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Obtention of a written informed consent.
* Patient with histologically proved cholangiocarcinoma ; histologic diagnosis must be proved by biliary brushing, bile cytology, endobiliary biopsy under Spyglass, or by EUS-FNA.
* Patient with Karnofsky score > 60， ECOG>level 2
* Patient capable of fill in the quality of life questionnaire
* For the first time treatment
* CT, MRCP, EUS and other examinations indicate that the tumor has locally infiltrated large blood vessels and cannot be surgically removed

Exclusion Criteria

* No written informed consent
* Patients under or already treated by radiotherapy or chemotherapy treatment for cholangiocarcinoma.
* Pregnant, parturient or breastfeeding women
* Serious abnormalities in liver and kidney function and coagulation function
* The ERCP guide wire cannot pass the stricture due to severe biliary stricture
* Merge with other malignant tumors
* Use other treatments that may affect the observation, such as radioactive particles or seed stent implantation, P53 injection, oral chemotherapy, interventional therapy, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
survival time | two years
  The period from endoscopic treatment to patient death or the last day of study

SECONDARY OUTCOMES:
Adverse events | one month
  Number of participants with adverse events; type, frequency and intensity of adverse events
Stent patency time | two years
  Take the stent placement as the starting point and the stent occlusion confirmed by ERCP as the end point. Record the time interval between the two point
Progression free survival | two years
  evaluate the survival time without disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.S, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laquiere A, Boustiere C, Leblanc S, Penaranda G, Desilets E, Prat F. Safety and feasibility of endoscopic biliary radiofrequency ablation treatment of extrahepatic cholangiocarcinoma. Surg Endosc. 2016 Mar;30(3):1242-8. doi: 10.1007/s00464-015-4322-7. Epub 2015 Jul 11. PMID 26162420
- [Background] Butros SR, Shenoy-Bhangle A, Mueller PR, Arellano RS. Radiofrequency ablation of intrahepatic cholangiocarcinoma: feasability, local tumor control, and long-term outcome. Clin Imaging. 2014 Jul-Aug;38(4):490-494. doi: 10.1016/j.clinimag.2014.01.013. Epub 2014 Feb 7. PMID 24637151
- [Background] Strand DS, Cosgrove ND, Patrie JT, Cox DG, Bauer TW, Adams RB, Mann JA, Sauer BG, Shami VM, Wang AY. ERCP-directed radiofrequency ablation and photodynamic therapy are associated with comparable survival in the treatment of unresectable cholangiocarcinoma. Gastrointest Endosc. 2014 Nov;80(5):794-804. doi: 10.1016/j.gie.2014.02.1030. Epub 2014 May 15. PMID 24836747